CLINICAL TRIAL: NCT02142478
Title: Theory-informed Evaluation of Two Delivery Approaches of a GP Exercise Referral Scheme
Brief Title: Evaluation of Two Different Delivery Approaches of a GP Exercise Referral Scheme
Status: Completed | Type: Observational
Sponsor: Liverpool John Moores University (Other)
Collaborators: Brock University (Other)
Responsible Party: Principal Investigator, Paula Watson, Lecturer/Senior Lecturer in Exercise and Health Psychology, Liverpool John Moores University
Other Study IDs: SPS-14-01; 14/YH/0160 (Other: National Research Ethics Service)
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Physical Activity
Keywords: physical activity; behaviour change; exercise referral; self-determination theory; mixed-method; evaluation; qualitative
MeSH Terms: conditions — Motor Activity | interventions — Health

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adapted scheme: Participants referred by their GP practices to Centre A will take part in the Adapted Exercise for Health (EFH) scheme.
  Interventions: Behavioral: Adapted Exercise for Health (EFH) scheme
- Standard scheme: Participants referred by their GP practices to Centre B will take part in the Standard Exercise for Health (EFH) scheme.
  Interventions: Behavioral: Standard Exercise for Health (EFH) scheme

INTERVENTIONS:
Behavioral: Adapted Exercise for Health (EFH) scheme — 12-week subsidised exercise programme at local authority-run leisure centres. Each participant receives a programme of activities tailored to their needs, based on a standard recommendation of two exercise sessions per week. In February 2012, Centre A introduced some changes to the EFH scheme as follows:
  * Pre-scheme meeting with a health trainer to help the patient decide if EFH is for them.
  * Participants offered specially tailored group classes (exclusive to EFH participants, e.g. low-impact circuits, Zumba) as well as access to the main gym.
  * Opportunities to attend daily.
  Although subsidised access to mainstream group classes and swim sessions (i.e. includes all leisure centre members) is also available, this option is not openly advertised on the adapted scheme.
  Groups: Adapted scheme
Behavioral: Standard Exercise for Health (EFH) scheme — 12-week subsidised exercise programme at local authority-run leisure centres. Each participant receives a programme of activities tailored to their needs, based on a standard recommendation of two exercise sessions per week.
  The scheme includes exclusive EFH gym sessions (i.e. includes EFH participants only) on two to three days of the week, plus subsidised access to mainstream group classes and swim sessions (i.e. includes all leisure centre members).
  Groups: Standard scheme

SUMMARY:
Physical activity (PA) benefits both physical and psychological health, yet the majority of UK adults are physically inactive. "Exercise for Health" (EFH) is a General Practitioner (GP) exercise referral scheme run in Liverpool for people who are inactive with a medical condition. Patients are referred by their GP practice, where they receive 12 weeks of subsidised exercise classes at their local leisure or community centre.

In 2012, one of the thirteen EFH centres (Centre A) introduced some changes to try and improve EFH at their centre. These changes included:

* a pre-scheme meeting with a health trainer, to help the patient decide if EFH is for them.
* exclusive classes (gym or activities) available daily for EFH participants (compared to gym only classes two or three times a week in other centres).

This non-randomised study will compare the effectiveness of the adapted EFH (Centre A) with standard EFH delivery (Centre B). All participants referred to centre A (n=100 approx) or centre B (n=100 approx) during the study period will be invited to take part. Changes in self-reported PA, PA self-efficacy and psychological wellbeing will be measured at the end of EFH (12 weeks) and at 12-month follow-up. A subsample of participants (n=15 from each centre) will take part in qualitative interviews to explore the factors that contribute to effectiveness.

A secondary aim is to explore psychological factors contributing to any differences between the two centres. Self-determination theory suggests that where participants feel they are offered choice, feel they are competent at exercise, and feel connected to people they exercise with, they will be more intrinsically motivated and more likely to continue exercising. Therefore it is hypothesised that participants attending the adapted EFH will be more motivated and more likely to continue exercising.

DETAILED DESCRIPTION:
This mixed-method observational study will compare the short- and long-term effectiveness of two different delivery approaches of an exercise referral scheme (Exercise for Health, EFH). As the intervention is already in widespread use randomisation is not feasible, therefore a case control design is adopted to compare the effectiveness of an adapted EFH scheme (delivered at centre A) with the standard EFH scheme (delivered at centre B). Centre B is selected as the comparison centre due to its similarity to centre A on socio-demographic markers (e.g. number of EFH referrals, socioeconomic make-up of local population).

Although the adapted scheme has not drawn overtly from Self-determination Theory (SDT), it is hypothesised that the adapted scheme promotes greater environmental support of SDT-based psychological needs for participants than the standard EFH scheme. Autonomy is promoted through the increased choice offered through daily sessions and the involvement of the patient in their decision whether to take up the scheme, competence is encouraged through the tailoring of classes to the ability of EFH participants and the opportunity to observe similar others, and relatedness is supported through the social assimilation of participants through regular group activities.

It is hypothesised that:

1. Both EFH delivery approaches will have beneficial effects on participants' self-reported PA, self-efficacy and psychological well-being post-intervention.
2. Participants attending the adapted scheme will perceive greater needs support, greater psychological needs satisfaction and more autonomous motivation during and post-intervention; will have higher adherence to EFH; will have higher leisure centre attendance from post-intervention to 12 months and report higher PA levels at 12 months.
3. Perceived needs support will predict psychological needs satisfaction during the intervention; psychological needs satisfaction during the intervention will predict autonomous motivation and psychological well-being post-intervention; post-intervention autonomous motivation will predict PA at 12 months and leisure centre attendance from post-intervention to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Individuals attending an EFH induction at centre A or centre B during the recruitment period (anticipated to be between May and July 2014).

Exclusion Criteria:

* Participants with an insufficient level of English language to understand the participant information sheet (in written or spoken format).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inactive adults (16+ years) who have, or are at risk of developing, a medical condition (e.g. hypertension, obesity, depression).
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in self-reported physical activity (PA) | Baseline, 12 weeks, 12 months
  Self-reported PA will be measured using the vigorous PA, moderate PA and walking items of the short version of the International Physical Activity Questionnaire (IPAQ). The short-IPAQ is a 7-day recall self-administered tool that measures intensity, frequency and duration of PA and provides a total estimate of energy expenditure. A total score of MET-minutes/week will be calculated according to the IPAQ scoring protocol, which is available to download from http://www.ipaq.ki.se/ipaq.htm

SECONDARY OUTCOMES:
Change in physical activity self-efficacy | Baseline, 12 weeks, 12 months
  A two-item measure of PA self-efficacy (SE) was developed to reflect the intervention aims. Item one measures self-efficacy to adhere to the Exercise for Health programme ("how confident are you that you can attend exercise sessions twice a week?"); item two measures self-efficacy to adhere to a physically active lifestyle in general ("how confident are you that you can be moderately physically active for at least 30 minutes on 5 days of the week?"). Participants are asked to rate their confidence on a scale of 0 (not at all confident) to 10 (extremely confident).
Change in psychological wellbeing | Baseline, 12 weeks, 12 months
  Psychological wellbeing will be measured using the Warwick-Edinburgh Mental Well-being Scale (WEMWBS). WEMWBS is a 14-item positively worded measure containing items related to psychological functioning (e.g. "I've been thinking clearly") and subjective well-being (e.g. "I've been feeling cheerful"). Participants are asked to rate on a likert scale of 1 (none of the time) to 5 (all of the time) how well each statement describes their experiences over the last two weeks.
Adherence to the Exercise for Health programme | Between baseline and 12 weeks
  Adherence will be expressed as a percentage of the recommended twice weekly leisure centre attendance over 12 weeks.
Post-intervention leisure centre attendance | Between 12 weeks and 12 months
  The number of occasions participants attend either gym sessions, classes or swim sessions between 12 weeks and 12 months will be obtained from computerised attendance records. Two measures will be taken: the absolute number of attendances (regardless of when these occur) and regularity of attendance (i.e. number of months in which participants attend at least once).

OTHER OUTCOMES:
Self-determination theory variables | 4 weeks, 12 weeks and 12 months
  Needs support (4 weeks and 12 weeks only) will be measured using a 15-item needs support (NS) tool that assesses participant perceptions of the extent to which their exercise referral instructors provide support for autonomy, structure (linked to competence) and involvement (linked to relatedness).
  Psychological needs satisfaction will be measured using the Psychological Need Satisfaction in Exercise Scale (PNSE). The PNSE is an 18-item tool designed to measure participants' perceived autonomy, competence and relatedness in an exercise context.
  Behavioural regulation of exercise will be measured using the revised Behavioural Regulation in Exercise Questionnaire (BREQ-2), which contains 19 items exploring reasons why people exercise. The scale includes items measuring amotivation, external regulation, introjected regulation, identified regulation and intrinsic motivation of exercise behaviour. Four additional items will be included to assess integrated regulation.
Qualitative interviews | 4 weeks and 12 months
  Qualitative interviews with a randomly-selected subsample of participants (15 per centre) will explore the following research questions:
  * What are the facilitators and barriers to exercise adoption for Exercise-for-Health (EFH) participants?
  * How acceptable is EFH to participants and how could it be improved?
  * How well do the processes of referral, induction and EFH activities at each centre support participants' perceived needs for autonomy, competence and relatedness?
  * What factors (EFH and individual) facilitate PA maintenance at 12 months?

CONTACTS AND LOCATIONS:
Overall Officials: Paula M Watson, PhD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom